CLINICAL TRIAL: NCT00354614
Title: Validation of the ApneaLink Sleep Screener in a Suspected Sleep Disordered Breathing Population
Brief Title: Validation of the ApneaLink Sleep Screener for Obstructive Sleep Apnea (OSA)
Status: Completed | Type: Observational
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Other Study IDs: CA-09-05
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: ApneaLink Sleep Screener — Device used to evaluate for the presence of OSA
  Other Names: AL

SUMMARY:
The primary endpoints for this study are that the AL validation will 1) achieve a sensitivity of greater than 80% for AHI values greater than or equal to 15, and 2) demonstrate a correlation coefficient of r=0.75 indicating strong correlation between the AHI of diagnostic PSG and AL.

DETAILED DESCRIPTION:
All subjects with suspected Sleep Disordered Breathing (SDB) scheduled for diagnostic polysomnography (PSG) will be invited to participate in the study to be tested to determine if they have Sleep Disordered Breathing (SDB), using the ApneaLink (AL) Sleep Screener. Subjects initially will be tested for SDB in the home environment. Following an AL home test, subjects will undergo a simultaneous, attended diagnostic polysomnography (PSG) sleep study and ApneaLink test for the purpose of confirming and comparing the results between diagnostic PSG and the AL device.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects ( greater than 18 years of age) of either gender or any race
* Suspected sleep disordered breathing
* Untreated sleep disordered breathing
* Willingness to use AL at home within 2 days of receipt and instruction on the AL
* Willingness to use AL at home and undergo PSG within 2 to 4 weeks of completing the at home AL test

Exclusion Criteria:

* Any subject requiring home oxygen therapy
* Any subject currently receiving positive airway pressure therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pts. with suspected OSA.
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2006-06; Primary Completion 2007-03 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J Strollo, MD, Principal Investigator — Associate Professor of medicine and Medical Director, UPMC Sleep Medicine
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Derived] Oktay B, Rice TB, Atwood CW Jr, Passero M Jr, Gupta N, Givelber R, Drumheller OJ, Houck P, Gordon N, Strollo PJ Jr. Evaluation of a single-channel portable monitor for the diagnosis of obstructive sleep apnea. J Clin Sleep Med. 2011 Aug 15;7(4):384-90. doi: 10.5664/JCSM.1196. PMID 21897775

RESULTS

PARTICIPANT FLOW:
Groups:
- Suspicion of Obstructive Sleep Apnea: Patients referred to a sleep clinic because of suspicion of obstructive sleep apnea underwent simultaneous polysomnography and ApneaLink testing
Period: Overall Study
Arm/Group | Suspicion of Obstructive Sleep Apnea
Started | 81
Completed | 53
Not Completed | 28
Not completed — Lack of Efficacy | 28

BASELINE CHARACTERISTICS:
Arm/Group | Suspicion of Obstructive Sleep Apnea
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 24
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 35.9 (9.1)

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity
Description: Comparison of sensitivity and specificity of ApneaLink to polysomnography with an apnea hypopnea index (AHI) cut-off of 15 or greater
Time Frame: Simultaneous single night recording
Measure: Number; unit: percentage
Arm/Group | Suspicion of Obstructive Sleep Apnea
Number analyzed (Participants) | 53
percentage
  Sensitivity | 79.0
  Specificity | 88.2

ADVERSE EVENTS:
Arm/Group | Suspicion of Obstructive Sleep Apnea
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No